CLINICAL TRIAL: NCT05778305
Title: Effect of Dexmedetomidine on Stress-induced Changes in Hemodynamics and Left Ventricular Function in Coronary Artery Bypass Graft Surgery Outcome
Brief Title: Effect of Dexmedetomidine on Left Ventricular Function in Coronary Artery Bypass Graft Surgery Outcome
Acronym: CABAG
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rania Maher Hussien, MD, Associate professor of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: FMASU MD283/2022
Record Dates: First submitted 2023-01-29; First posted 2023-03-21 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Effect of Drug in CABAG Patients
MeSH Terms: interventions — Dexmedetomidine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dexmedetomidine group (Active Comparator): patients will have loading Dexmedetomidine( 1ug/kg) over 10 minutes followed by continuous infusion of (0.5ug/kg/hr) from the initiation of anaesthesia up to extubation in the ICU. Patients will not be extubated until completely awake and have no sign of arrhythmias and bleeding
  Interventions: Drug: Dexmedetomidine
- control group (Placebo Comparator): patients will receive the same volume of 0.9% saline infusion as loading and maintenance infusion.
  Interventions: Other: normal saline

INTERVENTIONS:
Drug: Dexmedetomidine — a central sympatholytic drug
  Other Names: precedex
  Arms: Dexmedetomidine group
Other: normal saline — saline is given to control group
  Other Names: saline
  Arms: control group

SUMMARY:
50 patients of both sexes undergoing elective CABG surgery will be randomly divided into 2 groups, study group (Dex) group and control group (C) to determine the effect of dexmedetomidine on the peri-operative hemodynamic changes during CABG surgery.

DETAILED DESCRIPTION:
The effect of dexmedetomidine during CABG surgery is studied regarding Ventricular function, pre bypass and post bypass using the transoeophageal echo (TEE), post-operative by transthoracic echocardiography (TTE) on day of surgery and after extubation.

Incidence of intraoperative and post operative ischemia and arrhythmias using Electrocardiogram (ECG) as well as the length of ICU and hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* undergoing elective CABG surgery

Exclusion Criteria:

* Patient refusal

  * Dementia patients
  * Poor ventricular function with ejection fraction below 40%
  * Asthmatic patients
  * Uncontrolled diabetic patients with HbA1c above 8
  * Combined surgeries (CABG+ valves)
  * Emergency surgeries.
  * Pre-existing arrhythmia
  * Patients with renal impairment
  * Patients with hepatic impairment
  * Patients with heart block
  * Off-pump CABG

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-01-29 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Intra-operative ventricular function. | Intraoperative
  global systolic function Ejection Fraction by TEE intraoperative
post-operative ventricular function. | Up to 24 hours postoperative
  global systolic function Ejection Fraction by TTE postoperative

SECONDARY OUTCOMES:
hemodynamics | Immediate postoperative and up to 24 hours postoperative
  Heart Rate (beat/minute),
hemodynamics | Immediate postoperative and up to 24 hours postoperative
  Mean arterial blood pressure (mmHg)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Abassia, Egypt

IPD SHARING:
Plan to Share IPD: No